CLINICAL TRIAL: NCT04127851
Title: A Phase IV, Multicenter, Randomized, Single-blinded(Evaluator), Active-controlled, Parallel Study for Evaluating HA 0.15% Compared With Cyclosporine 0.05%, and Efficacy of Combination Therapy in Moderate to Severe Dry Eye Disease Patients
Brief Title: Evaluating HA 0.15% Compared With Cyclosporine 0.05%, and Efficacy of Combination Therapy in Dry Eye Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJO-018
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins; Standard of Care; MCC protocol

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Single-blind Study for Evaluating the Efficacy of HA 0.15% Compared with Cyclosporine 0.05% in Moderate to Severe Dry Eye Syndrome
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium Hyaluronate 0.15% mono-therapy (Experimental): HA 0.15% group was treated with HA 0.15% six times daily for 12 weeks
  Interventions: Drug: TJO-018 (HA 0.15%)
- Cyclosporin 0.05% + carboxymethylcellulose (CMC) 0.5% (standard therapy) (Active Comparator): CsA 0.05% + CMC 0.5% group was treated with CsA 0.05% two times daily and CMC 0.5% two ~ six times daily for 12 weeks.
  Interventions: Drug: Cyclosporine Ophthalmic Emulsion 0.05% standard therapy (CMC 0.5% add)
- HA 0.15% + CsA 0.05% (combination therapy) (Other): HA 0.15% + CsA 0.05% group was treated with HA 0.15% six times daily and CsA 0.05% twice daily for 12 weeks.
  Interventions: Drug: TJO-018 (HA 0.15%) + Cyclosporine Ophthalmic Emulsion 0.05%

INTERVENTIONS:
Drug: TJO-018 (HA 0.15%) — TJO-018 / one drop / 6 times daily in both eyes
  Arms: Sodium Hyaluronate 0.15% mono-therapy
Drug: Cyclosporine Ophthalmic Emulsion 0.05% standard therapy (CMC 0.5% add) — Cyclosporine / one drop / twice daily in both eyes carboxymethylcellulose (CMC) / one drop / two~six times daily in both eyes
  Arms: Cyclosporin 0.05% + carboxymethylcellulose (CMC) 0.5% (standard therapy)
Drug: TJO-018 (HA 0.15%) + Cyclosporine Ophthalmic Emulsion 0.05% — TJO-018 (HA0.15%)/ one drop 6 times daily in both eyes Cyclosporine 0.05% /one drop twice daily in both eyes
  Arms: HA 0.15% + CsA 0.05% (combination therapy)

SUMMARY:
In patients with moderate to severe dry eye syndrome, the test drug (HA 0.15% eye drop) or the control drug (cyclosporin 0.05% eye drop) is administered for 12 weeks, and the corneal staining of each group would be evaluated. The study objective is to demonstrate that the test drug is not clinically inferior to the control drug.

Furthermore, the efficacy of combination therapy would be evaluated through exploratory combination therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Moderate to Severe Dry Eye Disease Patients
* Written informed consent to participate in the trial

Exclusion Criteria:

* Any laser or ocular surgery within 2 months prior screening
* Use of contact lenses
* Any condition limiting patient's ability to participate in the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Corneal Staining Score at Week 12 | Baseline and Week 12
  After 12 weeks of administration of the drugs compare the therapeutic effectiveness between control drug and trial drug evaluated as the corneal staining score change.
  * Scale: "Oxford grading system" that divides into six groups according to severity from 0 (absent) to 5 (severe).
  * The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change From Baseline in Corneal Staining Score at Week 4 and Week 8 | Baseline, Week 4 and Week 8
  After 4, 8 weeks of administration of the drugs compare the therapeutic effectiveness between control drug and trial drug evaluated as the corneal staining score change.
  * Scale: "Oxford grading system" that divides into six groups according to severity from 0 (absent) to 5 (severe).
  * The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, South Korea